CLINICAL TRIAL: NCT03419429
Title: The Use of Simvastatin Gel With Perforated Resorbable Membranes in the Treatment of Intrabony Defects in Chronic Periodontitis Patients (Clinical and Biochemical Study)
Brief Title: Simvastatin Gel With Perforated Resorbable Membranes in Treatment of Intrabony Defects in Chronic Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dalia Rasheed Issa, Associate lecturer of oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-RECD 12165332
Record Dates: First submitted 2018-01-17; First posted 2018-02-05 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Chronic Periodontitis
Keywords: Guided tissue membranes; EDTA; Simvastatin
MeSH Terms: conditions — Chronic Periodontitis | interventions — Simvastatin; Edetic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Simvastatin/Occlusive membrane (Experimental): open flap procedure, 1.2%simvastatin gel applied and covering the defect with resorbable collagen occlusive membrane .
  Interventions: Drug: Simvastatin; Device: Occlusive membrane
- Simvastatin/perforated membrane (Experimental): open flap procedure, 1.2% simvastatin gel and covering the defect with resorbable collagen modified perforated membrane.
  Interventions: Drug: Simvastatin; Device: Modified perforated membrane
- EDTA/Simvastatin/Occlusive membrane (Experimental): open flap procedure, 24% EDTA root surface etching,1.2% simvastatin gel and then coverage of the defect with occlusive membrane.
  Interventions: Drug: Simvastatin; Other: EDTA; Device: Occlusive membrane
- EDTA/Simvastatin/perforated membrane (Experimental): open flap procedure, 24% EDTA root surface etching, 1.2% simvastatin gel and then coverage of the defect with modified perforated membrane.
  Interventions: Drug: Simvastatin; Other: EDTA; Device: Modified perforated membrane

INTERVENTIONS:
Drug: Simvastatin — Simvastatin is a drug used orally for treatment of hypercholesterolemia. It assists in bone regeneration and has anti-inflammatory effect when applied locally in intrabony defects for periodontal therapy.
Other: EDTA — EDTA is a demineralizing agent used for root surface conditioning.
  Other Names: Ethylenediaminetetraacitic acid
  Arms: EDTA/Simvastatin/Occlusive membrane; EDTA/Simvastatin/perforated membrane
Device: Occlusive membrane — Occlusive membrane is the traditional collagen resorbable membrane used in guided tissue regeneration.
  Other Names: Resorb resodont forte
  Arms: EDTA/Simvastatin/Occlusive membrane; Simvastatin/Occlusive membrane
Device: Modified perforated membrane — Modified perforated membrane is the traditional collagen resorbable membrane but modified to be perforated. It is used in guided tissue regeneration
  Other Names: Resorb resodont forte
  Arms: EDTA/Simvastatin/perforated membrane; Simvastatin/perforated membrane

SUMMARY:
Modified perforated membrane (MPM) is considered as a modality that could enable participation of periosteal cells and gingival stem cells which could improve the outcomes of guided tissue regeneration more than the use of the traditional occlusive membrane (OM). Simvastatin (SMV) modulates bone formation by increasing the expression of bone morphogenetic protein 2 and angiogenesis. Ethylenediaminetetraacitic acid (EDTA) found to be effective as low ph etchant for smear layer removal and exposing root surface collagen. The investigators compared the clinical and radiographic outcome of SMV gel combined with MPM to SMV gel combined with OM with and without an associated EDTA gel root surface etching for improving bone regeneration in intrabony defects in chronic periodontitis patients. Moreover, evaluation of SMV gingival crevicular fluid (GCF) levels availability for 30 days in cases with and without EDTA root surface etching was performed.

DETAILED DESCRIPTION:
Forty patients with 40 intrabony defects having chronic periodontitis were randomly assigned into four equal groups to receive open flap procedure, 1.2% SMV gel and covering the defect with OM (Group I), open flap procedure, 1.2% SMV gel and covering the defect with MPM (Group II), open flap procedure, 24% EDTA root surface etching,1.2% SMV gel and then coverage of the defect by OM (Goup III), or open flap procedure, 24% EDTA root surface etching, 1.2% SMV gel and then coverage of the defect by MPM (Group IV). Plaque index, gingival index,probing pocket depth, clinical attachment level, defect base level, crestal bone level, and radiodensitometric measurements were measured at baseline and reassessed at 6 and 9 months after therapy. Additionally, GCF was collected from group I, II, III and IV at 1,7,14, 21, and 30 days in order to evaluate SMV availability and the effect of EDTA root surface etching on its availability using High-performance liquid chromatography(HPLC).

ELIGIBILITY:
Inclusion Criteria:

* Patients were all healthy and free from any systemic disease.
* No history of antibiotic therapy or periodontal treatment for at least six months preceding the study.
* Patients were willing and able to return for multiple follow up visits.
* Periodontal defects with

  1. Probing depth > 5 mm.
  2. Clinical attachment loss >4 mm.
  3. Standardized radiographic evidence of interproximal intrabony defect using periapical radiograph.
* Good level of oral hygiene (plaque and gingival indices score after initial phase therapy should be less than one).

Exclusion Criteria:

* Pregnancy, lactation for female patients.
* Smokers, alcoholics and those receiving any medication that could affect healing of soft tissue and bone as steroids and cyclosporines.
* History of allergic reaction to the medications used.
* Vulnerable groups and handicapped.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth | Baseline to 9 months
  Probing pocket depth was measured from the free gingival margin to the base of the pocket from baseline to 6 months and 9 months
Clinical attachment level | Baseline to 9 months
  Clinical attachment level was measured from the cementoenamel junction to the base of the pocket from baseline to 6 months and 9 months
Plaque index | Baseline to 9 months
  Plaque index was measured from baseline to 6 months and 9 months
Gingival index | Baseline to 9 months
  Gingival index was measured from baseline to 6 months and 9 months
Linear measurements | Baseline to 9 months
  Linear measurements were measured using Digora software from baseline to 6 months and 9 months
Radiodensitometric measurements | Baseline to 9 months
  Bone density was measured using Digora software from baseline to 6 months and 9 months

SECONDARY OUTCOMES:
Simvastatin gingival crevicular fluid levels | Day 1, 7, 14, 21 and 30
  Simvastatin gingival crevicular fluid levels availability in cases with and without EDTA root surface etching using HPLC at day 1, 7, 14, 21,and 30

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Y Gamal, Professor, Study Director — Faculty of dentistry- Ain Shams University